# **Informed Consent Form**

Study Title: Mobile Evidence-Based Smoking Cessation for Veterans Living With HIV (MESH)

NCT Number: NCT04135937

Document Date: 3/31/2021

| Department of Veterans Affairs | Research Informed Consent Form | | |
|---|---|---|---|
| Department of Veterans Anans | Version Date: 3/31/2021 | L | |
| Participant Name: | | Date: | |
| Study Title: Smoking Cessation Treatment Preferences among Veteran Smokers Living with HIV | | | |
| Principal Investigator: Sarah Wilson, PhD | | VAHCS: | Durham VAMC |

#### **OVERVIEW AND KEY INFORMATION**

Please read this form carefully. You are being asked to participate in this research study because you may have current HIV infection and tobacco use. This study is voluntary and will include only people who choose to take part. Ask your study doctor or study staff to discuss this consent with you, please ask him/her to explain any words or information that you do not understand. It is important that you understand the information on this form.

The purpose of this study is to learn more about ways to help veterans living with HIV quit smoking.

Your participation in this study will involve smoking cessation medication, at least 5 counseling sessions, and smoking cessation supporting text messaging (if you have a cell phone and are willing to receive messages). You will also be asked to complete questionnaires, interviews, and breath and saliva samples before and after treatment.

The greatest risks of this study involve experiencing smoking withdrawal symptoms when you quit smoking. Quitting smoking will cause nicotine withdrawal that may lead to headaches, nausea, irritability, weight gain, difficulty concentrating, poor sleep, increased appetite, anxious or depressed mood, and craving for cigarettes.

#### WHY IS THIS STUDY BEING DONE?

The study is being done to learn more about ways to help veterans living with HIV quit smoking. You are being asked to participate in this research study because you may currently meet criteria, including HIV infection and current tobacco use. This study is being run by Dr. Sarah Wilson.

#### HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY

Approximately 15 people will be enrolled in this study at the Durham VA Health Care System.

| Subject Identification (Last, First, Middle Initial) | IRB Approval Date |
|---|---|
| | DVAHCS Template Version Date: 12/20/18 |

| Department of Veterans Affairs | Research Informed Consent Form | | |
|---|---|---|---|
| Department of Veteralis Allans | Version Date: 3/31/2021 | L | |
| articipant Name: | | Date: | |
| Study Title: Smoking Cessation Treatment Preferences among Veteran Smokers Living with HIV | | | |
| Principal Investigator: Sarah Wilson, PhD | | VAHCS: [ | Ourham VAMC |

#### HOW LONG WILL I BE IN THIS STUDY?

Your participation in this study will last about 6 months, but most of your work in the study happens during the first two months or so.

#### WHAT IS INVOLVED IN THIS STUDY?

If you agree to participate in this research study you will be asked to sign and date this consent form. In the baseline session (Session 0), we will ask you a series of questions related to your mood, beliefs, medical history, quality of life, substance use, and your smoking history. During the COVID-19 pandemic, this session and others may occur remotely using VA Video Connect or another approved platform. After the pandemic, you will be asked to visit our lab. You will be asked to provide a breath sample so that we can measure the carbon monoxide (CO) in your breath, as well as a saliva sample. These are measures of smoking. Because we are interested in learning about how stopping smoking affects HIV and AIDS among Veterans, we will review your computerized medical record, collecting some information about your health, including laboratory results, diagnoses, and medications.

You will then be scheduled for counseling session 1 with a stop smoking counselor within 7 days of study enrollment. Counseling sessions will be individually tailored to your preferences and treatment experience. This will occur in person at the Durham VA Health Care System. For subsequent counseling sessions, you will be offered the choice of whether to complete counseling sessions using a personal telephone, a personal digital device (i.e., tablet, laptop, or desktop computer with webcam), or a VA-issued digital device (i.e., 4G-enabled tablet with webcam). If you request to use a VA-issued personal digital device, we will place a consult to Prosthetics Service to get you the device. If you use a VA device, your counseling sessions may occur via VA Video Connect or another approved platform.

Counseling sessions are designed to help you get ready to make a quit attempt, make a quit attempt, and avoid relapse to smoking. Your treatment sessions may include topics like depression, posttraumatic stress disorder (PTSD), alcohol use, pain, weight gain, medications for helping stop smoking, and other topics. Each counseling session will last 30 to 60 minutes. You will participate in at least 5 sessions. These sessions will be audio recorded for fidelity purposes. Part of this treatment may involve consulting with your other health care providers at VA. We will not consult with any health care provider without your knowledge and assent. If we do consult with one of your VA health

| Department of Veterans Affairs | Research Informed Consent Form | | |
|---|---|---|---|
| Department of veteralis Arians | Version Date: 3/31/2021 | L | |
| Participant Name: | I | | Date: |
| Study Title: Smoking Cessation Treatment Preferences among Veteran Smokers Living with HIV | | | |
| Principal Investigator: Sarah Wilson, PhD | | VAHCS: [ | Durham VAMC |

care providers, treatment-relevant health information may be recorded in the electronic medical record.

At counseling Session 1, your counselor will ask you questions regarding smoking cessation medication preferences and contraindications. The staff member will also review your electronic medical record to see if you have any contraindications to medication use.

At counseling session 1 we will ask you to sign up for personalized text messaging support. This text support will be provided using a program called SmokefreeVET or the VA Annie app. SmokefreeVET is a national online smoking cessation program that provides supportive text messages to Veterans who are interested in quitting smoking. You can opt out of messaging at any time. Annie is an automated, short message service (SMS) text message system designed to promote Veteran self-care. It is not designed to allow you to contact a provider in a medical emergency. If you have a working cell phone and are willing to receive SMS text messages, we will send you messages starting after Session 1 and extending through 6 months after you make a quit attempt. We will tailor the messages to you receive based on your preferences on topic, type, and frequency. You can opt out of messaging at any point.

At Session 3 (1 week after your quit-smoking date), you will be asked several questions designed to help us further personalize your smoking cessation treatment. Your information will be entered into a computerized system that will design a personal treatment. Your treatment may include additional counseling sessions or taking medications for helping you stop. If the computer system recommends taking medications, we will send these recommendations to your ID Clinic team. All prescriptions will be managed as part of routine clinical care by your VA healthcare providers, who may choose to follow or not to follow our recommendations.

You will asked to participate in other study sessions immediately following your end of counseling, and then 3 months and 6 months after you started treatment for follow-up sessions. During these return visits you will complete measurements and be interviewed. The post-treatment interview will include questions regarding strengths and weaknesses of the intervention as well as suggestions for ways to improve the overall treatment approach. This interview will be audio-recorded. We will pay you \$50 for participating in the interview. During the COVID-19 pandemic, we will mail you a CO monitor at these three time points. You will be asked to provide a breath sample during a video call.

| | Research Informed | Consont Form |
|---|---|---|
| Department of Veterans Affairs | Version Date: 3/31/2021 | |
| Participant Name: | | Date: |
| Study Title: Smoking Cessation Treatment Preferences am | nong Veteran Smokers Living with | HIV |
| Principal Investigator: Sarah Wilson, PhD | | VAHCS: Durham VAM |
| You will then return the CO monitor to us by mail, equipment. After the pandemic, if it is safe to do so samples in person at these times points. | | |
| The VA has recently approved use of an email progregarding study procedures. If you are comfortable questionnaires, or other study messages via email, coordinator or your study therapist. | e receiving appointment remind | ders, study |
| Your data may be stored and used for future studie identifiable private information, such as your name | | • |
| Future Use of Data and Contact for For If you consent to participate in this research study, you in the future. We will store this contact inform database called "Contact Database." This database used to determine if you may be eligible for future Research Laboratory and to contact you about parrelated to smoking, posttraumatic stress disorder (Your choice to give permission to be re-contacted not affect your enrollment in the current study. If you we will not contact you in the future about other standards. | we will collect information about the stored at the DVAHCS. This is stored at the DVAHCS. This is studies run in the Traumatic Sticipation. These future studies (PTSD), and trauma. This permit or not to give permission to be you do not wish for us to keep | w results in a information will be tress and Health include studies ssion is optional. re-contacted will |
| I agree to be re-contacted about participati | ing in future research studies: [ | Yes No |
| Only if you grant permission, data collected from y entered into a large database called "Trauma Data Data will not include any identifying information, a | base." This data will be used fo | or future research. |

I agree to future use of my data:  $\square$  Yes  $\square$  No

| Department of Veterans Affairs | Research Informed Consent Form | | |
|---|---|---|---|
| | Version Date: 3/31/2021 Page 5 | | |
| Participant Name: | | | Date: |
| Study Title: Smoking Cessation Treatment Preferences among Veteran Smokers Living with HIV | | | |
| Principal Investigator: Sarah Wilson, PhD | | VAHCS: [ | Ourham VAMC |

#### WHAT ARE THE RISKS AND DISCOMFORTS OF PARTICIPATING IN THIS RESEARCH STUDY?

There are some risks to participating in the study. First, you may have some discomfort related to quitting smoking. Quitting smoking will cause nicotine withdrawal that may lead to headaches, nausea, irritability, weight gain, difficulty concentrating, poor sleep, increased appetite, anxious or depressed mood, and craving for cigarettes. If your physician prescribes medications to help you stop smoking based on our recommendation, there may be side effects associated with those medications. Your physician and/or the VA pharmacist will inform you about these potential side effects. There is the potential risk of loss of confidentiality. Every effort will be made to keep your information confidential; however, this cannot be guaranteed. Some questions asked as part of this study may make you feel uncomfortable or increase distress. This discomfort or increased distress is usually temporary and well tolerated. You do not have to answer questions and you can take a break at any time. You can call the study team at any time if you experience any discomfort related to the research.

If you choose to take part in this study, you are at risk for the following risks or side effects. You should discuss these with your study doctor.

#### WILL I BENEFIT FROM TAKING PART IN THIS RESEARCH STUDY?

You may not personally benefit from taking part in this study, but your participation may lead to knowledge that will help people in the future. You may benefit from stopping smoking, but this benefit is not guaranteed to you.

#### WHAT OTHER OPTIONS OR ALTERNATIVES DO I HAVE?

Taking part in this study is your choice. You may choose to not participate. If you choose not to participate, you may be eligible for usual VA smoking cessation treatments. The study team will talk to you about what those treatments are like and how to enroll.

#### HOW WILL MY RESEARCH DATA BE PROTECTED AND SECURED?

Your information used for this study will be kept confidential as required by law. The results of this study may be used for scientific purposes or for publication, but these results will not include any information that would identify you. Your identity will not be disclosed without your consent, or

| Department of Veterans Affairs | Research Informed Consent Form | | |
|---|---|---|---|
| Department of Veteralis Allans | Version Date: 3/31/2021 | Ĺ | |
| Participant Name: | Da | | Date: |
| Study Title: Smoking Cessation Treatment Preferences among Veteran Smokers Living with HIV | | | |
| Principal Investigator: Sarah Wilson, PhD | | VAHCS: [ | Durham VAMC |

unless required by law. Your research records will be maintained and destroyed according to VHA records retention requirements.

All study data will be kept in a secured file to which only study team members will have access. Hard copy paper records (that is, any forms you sign) will be stored in a locked filing cabinet in the study coordinator's locked office, within this research lab at the Durham Veteran's Affairs Health Care System. Information collected during your sessions will be entered into a computerized database. This database is stored on a VA secured computer server that is password-protected, and only accessible by Dr. Wilson and her study staff. An audio recording of your interview will be stored temporarily on the audio recorder, which is kept in our research laboratory's office in a locked filing cabinet. The recording will be moved to a VA secured computer server that is password-protected. From there, they may be moved to an encrypted DVD that is password-protected. Only study staff members have access to the passwords that protect your information.

Access to data stored at the Durham VA Health Care System will be limited to a small number of study team members who have been trained to preserve participant confidentiality. The key linking code numbers and identifying information will be kept in a locked office in the Durham VA, and will be maintained on password-protected computers behind the VA firewall on the VA secured server.

If you are asked to provide a saliva sample, the sample you provide will be mailed to an outside laboratory to be analyzed. This sample will be identified only with a study identification number.

Your research records may be reviewed by Durham VA staff who are responsible for the safe conduct of this research. We may also provide your research records to federal agencies such as the Office for Human Research Protections (OHRP), the VA Office of the Inspector General (OIG), and the Office of Research Oversight (ORO). We will not share any information with these groups outside the VHA unless they agree to keep the information confidential and use it only for the purposes related to the study. Any information shared with these outside groups may no longer be protected under federal law. These groups may disclose your information to other groups. If the sponsor receives identified information, it is then the sponsor, and not the VA, who is responsible for the security of the information.

| Department of Veterans Affairs | Research Informed Consent Form | | |
|---|---|---|---|
| Department of Veterans Analis | Version Date: 3/31/2021 | 1 | |
| Participant Name: | | Date: | |
| Study Title: Smoking Cessation Treatment Preferences among Veteran Smokers Living with HIV | | | |
| Principal Investigator: Sarah Wilson, PhD | | VAHCS: [ | Ourham VAMC |

#### DOES PARTICIPATION IN THIS RESEARCH STUDY COST ANYTHING?

There will be no costs to you for any of the research treatment or research testing done as part of this research study. Some Veterans are required to pay co-payments for medical care and services provided by VA. These co-payment requirements will continue to apply to medical care and services provided by VA that are not part of this study. If your physician decides to prescribe you medications that are recommended by our study team, you may be responsible for co-payments for those medications.

# WILL I RECEIVE ANY COMPENSATION (MONEY OR OTHER) FOR TAKING PART IN THIS RESEARCH STUDY?

You will be reimbursed up to \$350 for your participation in this study. You will be compensated \$50 for each of the 4 data collection visits (baseline, post-treatment, 3-month follow-up, and 6-month follow-up). You may be paid \$50 each time you return the CO monitor if you are loaned one because you cannot attend an in-person visit (up to \$150).

Money that you receive for participating in research is considered taxable income per Internal Revenue Service (IRS) regulations. The money may be reported to the IRS and you may receive an IRS Form 1099.

### WHAT WILL HAPPEN IF I AM INJURED WHILE PARTICIPATING IN THE RESEARCH STUDY?

The VA will provide necessary medical treatment should you be injured by being in this study. You will be treated for the injury at no cost to you. This care may be provided by the Durham VAHCS or arrangements may be made for contracted care at another facility. Every reasonable safety measure will be taken to protect your well-being. You have not released this institution from liability for negligence. In case of research related injury resulting from this study, you should contact your study team. If you have questions about compensation and medical treatment for any study related injuries, you can call the medical administration service at this VA Medical Center at 919-286-6957.

| Department of Veterans Affairs | Research Informed Consent Form | | |
|---|---|---|---|
| Department of Veterans Analis | Version Date: 3/31/2021 | L | |
| Participant Name: | nt Name: | | Date: |
| Study Title: Smoking Cessation Treatment Preferences among Veteran Smokers Living with HIV | | | |
| Principal Investigator: Sarah Wilson, PhD | | VAHCS: [ | Durham VAMC |

### WHAT ARE MY RIGHTS TO DECLINE PARTICIPATION OR WITHDRAW FROM THE STUDY?

You can choose to not be in this study, or, if you agree to be in the study, you can withdraw at any time. If you withdraw from the study, no new data about you will be collected for study purposes. We will keep and use the data that we already collected before you withdrew your consent.

If you choose to not be in the study or if you withdraw from the study, there will be no penalty or loss of any benefits to which you are otherwise entitled. This will not affect your relationship with or treatment by the Veterans Health Administration (VHA) or your rights as a VHA patient. You will still receive all the medical care and benefits for which you are otherwise eligible.

<u>Withdrawal of Data for Future Use</u> If you agree to allow your data with information that would link the data to you to be kept for future research or for re-contacting, you can change your mind at any time. To withdraw your data, contact Dr. Sarah Wilson in writing and let him/her know you are withdrawing permission for your identifiable data to be used for future research. Dr. Wilson's mailing address is:

Durham VA Health Care System Attn: 152, Dr. Sarah Wilson 508 Fulton Street Durham, NC 27705

If your identifying information, such as your name or medical record number, are removed, we will no longer be able to identify and withdraw your data.

#### ARE THERE REASONS THAT MY RESEARCH PARTICIPATION MAY END EARLY?

Dr. Wilson may take you out of the study without your consent for one or more of the following reasons: 1) failure to follow instructions of investigator and/or study staff, 2) inability to complete study procedures, or 3) the study staff cannot reach you by telephone after multiple attempts.

We will tell you about new information that may affect your health, condition, welfare, or willingness to participate in this study.

| Department of Veterans Affairs | Research Informed Consent Form | | |
|---|---|---|---|
| Department of Veteralis Arians | Version Date: 3/31/2021 | L | |
| Participant Name: | | Date: | |
| Study Title: Smoking Cessation Treatment Preferences among Veteran Smokers Living with HIV | | | |
| Principal Investigator: Sarah Wilson, PhD | | VAHCS: [ | Durham VAMC |

#### WILL THE RESULTS OF THIS RESEARCH STUDY BE SHARED WITH ME?

We do not routinely send out results of the research study. However, if you would like to receive copies of any journal articles that are written using the data we gather during this study, please tell the study coordinator. He/she will make note, and send you a copy of any article about this study.

# DO ANY OF THE RESEARCHERS HAVE A FINANCIAL INTEREST RELATED TO THIS RESEARCH STUDY?

This study is funded by the Department of Veterans Affairs, and portions of the study staff members' salaries are paid by this study.

# WHERE CAN I FIND OTHER INFORMATION ABOUT THIS RESEARCH STUDY?

A description of this clinical trial will be available on *http://www.ClinicalTrials.gov*, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# WHO DO I CONTACT IF I HAVE QUESTIONS OR CONCERNS ABOUT THE RESEARCH STUDY?

If you have questions about the research or need to talk to the study team, you can contact Dr. Wilson at 919-808-5891during regular business hours or after hours. If you have questions about the research or your rights as a research participant, would like to obtain information, offer input, or have other concerns or complaints, you may contact the administrative officer of the research service at (919) 286-0411, extension 177632. If you would like to check that this study is approved by the Durham VAHCS's Institutional Review Board, please call the research office at (919) 286-6926 or (888) 878-6890, extension 176926.

| Department of Veterans Affairs | Research Informed Consent Form | |
|---|---|---|
| Department of Veterans Arians | Version Date: 3/31/2021 | Page 10 of |
| Participant Name: | | Date: |
| Study Title: Smoking Cessation Treatment Preferences a | mong Veteran Smokers Living with | HIV |
| Principal Investigator: Sarah Wilson, PhD | | VAHCS: Durham VAM |
| AFFIRMATION FROM PARTICIPANT I have read this form or it has been read to me. I explained to me, and I voluntarily consent to pare explanation of what the study is about and how disclosure of my identifiable information as described this consent form. | rticipate in this study. I have rec<br>and why it is being done. I auth | ceived an<br>norize the use and |

Date

Date

Signature of Participant

Signature of Person Obtaining Consent